CLINICAL TRIAL: NCT03572751
Title: Suitability of Unobtrusive Bed Monitoring and Wrist-worn Heart Rate Monitor for Patient Monitoring
Acronym: BedMon
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R17027
Record Dates: First submitted 2018-03-26; First posted 2018-06-28 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Arrhythmia; Hemorrhage; Septic Shock; Consciousness, Loss of; Sleep
Keywords: Sensor; Wearable
MeSH Terms: conditions — Arrhythmias, Cardiac; Hemorrhage; Shock, Septic; Unconsciousness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vascular surgical patients: Patient subjects are recruited from patients referred for vascular surgical procedure in Tampere University Hospital.
  Bed-, wrist- and ECG-sensor monitoring
  Interventions: Diagnostic Test: Bed-, wrist- and ECG-sensor monitoring
- Healthy volunteers: Healthy volunteer subjects will be recruited mainly from the students of Tampere University of Technology.
  Bed-, wrist- and ECG-sensor monitoring
  Interventions: Diagnostic Test: Bed-, wrist- and ECG-sensor monitoring

INTERVENTIONS:
Diagnostic Test: Bed-, wrist- and ECG-sensor monitoring — Bed-, wrist- and ECG-sensor monitoring

SUMMARY:
Novel technology enables it to monitor noninvasively the vital signs of a patient. Such a monitoring is immediately required to improve patient safety and to reduce hospital readmissions. In this study, novel bed- and wearable sensors are studied for this purpose.

DETAILED DESCRIPTION:
Unobtrusive bed monitoring devices have gained popularity in the area of voluntary sleep quality monitoring for wellness purposes. Most of these devices rely on the measurement of ballistocardiographic forces caused by the acceleration of blood when the heart pumps it to aorta, forces caused by respiration movements and other movements of the person being monitored. A thin film-type force sensor placed under the bed mattress, between the matrices or under the bed sheet is often used for measuring these forces. While proven to provide adequate reliability and accuracy for wellness monitoring of healthy people, unobtrusive bed monitoring solutions have not yet been widely deployed in hospital patient monitoring even though there would be much use for such technology e.g. in regular hospital wards where currently the amount of patient monitoring is very limited.

If proven operational in this application, bed monitoring technology would provide tremendous benefits in both clinical and home monitoring scenarios. Wrist worn pulse plethysmography (PPG) devices have increased their popularity as heart rate monitors, referred as optical heart rate monitors (OHR) for sports and wellness in recent years and their ability to measure average heart rate during movement and beat-to-beat heart rate while at rest accurately with healthy people has been shown.

The objective of the study is to collect ECG and movement data measured with a wearable ECG monitor and simultaneously record data with unobtrusive bed sensor and wrist worn PPG device. Data recorded with the bed and wrist sensors and vital parameters calculated from that or provided by the monitoring devices directly will be compared with the reference.

The purpose of the study is to gain knowledge about the feasibility of unobtrusive bed and wrist monitoring devices for patient monitoring. The collected data will directly provide information on the accuracy of the current algorithms of the monitors. Besides this evaluation, the collected data will be used in developing new algorithms for detection of cardiac problems.

The study includes collection of data from vascular patients referred to surgical operation in Tampere University Hospital. Data collection takes place at vascular surgical ward where one dedicated research bed is equipped with bed monitoring devices. Another group of subjects is formed by healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age>50
* Indication for operation: peripheral arterial bypass and/or endarterectomy, aortic surgery, carotid surgery
* Volunteering

Exclusion Criteria:

* Pacemaker
* Denial

Ages: 50 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caucasian
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy and precision of heart rate (1/s) measurement by a bed sensor | 24 hours
  Comparison of bed sensor derived heart rate with ECG reference to determine accuracy and precision of heart rate measurement by a bed sensor
Accuracy and precision of heart rate variability (ms) measurement by a bed sensor | 24 hours
  Comparison of bed sensor derived heart rate variability with ECG reference
Accuracy and precision of respiratory rate (1/min) measurement by a bed sensor | 24 hours
  Comparison of bed sensor derived respiratory rate measurement with accelerometer derived reference
Accuracy and precision of body movement detection | 24 hours
  Comparison of bed sensor derived body movement with accelerometer derived reference

SECONDARY OUTCOMES:
Duration of light sleep | 24 hours
  Measurement of light sleep duration by bed-worn sensor
Duration of rapid eye movement (REM) sleep | 24 hours
  Measurement of REM sleep duration by bed-worn sensor
Duration of deep sleep | 24 hours
  Measurement of deep sleep duration by bed-worn sensor

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No